CLINICAL TRIAL: NCT05357222
Title: Impact of Vocal Fold Stretching Exercise on Pitch Range and Phonation Stability
Brief Title: Straw Phonation Exercise Program for Pitch Extension
Acronym: SOVT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Lynn Maxfield, Research Scientist, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB_00141650; R01DC018280 (NIH)
Record Dates: First submitted 2021-05-10; First posted 2022-05-02 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Voice Fatigue; Voice Disorders; Voice Hoarseness
MeSH Terms: conditions — Voice Disorders; Hoarseness

STUDY DESIGN:
Intervention Model Description: Participants will be grouped based on their daily vocal usage (i.e. vocal user (4+ hours of speaking per day) or low vocal user (less than 4 hours per day). Both groups will be given a series of vocal stretching exercises that will be completed through a 2mm diameter straw.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Straw Phonation (Experimental): Participants will undergo one session of voice habilitation via a straw phonation exercise protocol. This protocol has been extensively studied and validated in the largest randomized clinical trial in voice therapy by our team.
  Interventions: Behavioral: Straw phontion

INTERVENTIONS:
Behavioral: Straw phontion — Pitch Glides: (1 minute) Vocalize through the straw starting from as low as possible to as high as possible. As the participant you will want to get as much as your vocal range as possible. But, don't let the voice get growly at the bottom or press it into a painful range at the top.
  2. Accents: (1 minute) Vocalize progressive little hills or accents. It sounds like a revving engine of the car.
  3. Song: (1 minute) Pick a favorite song and vocalize it through the straw. Examples: National Anthem, Happy Birthday, Mary had a Little Lamb. These are great songs because they have a range of pitches and one can build some accents in, as well.
  4. Reading passage: (1 minute) Vocalize a reading passage through the straw. Be as dramatic as possible, using a lot of inflection.
  Other Names: Semi-occluded vocal tract exercises, flow resistant tube

SUMMARY:
To investigate the change in fundamental frequency range and vocal fold stability achievable with vocal fold stretching exercise in human populations with high and low vocal activity

DETAILED DESCRIPTION:
The vocal ligament is part of the layered structure of the vocal fold. It is a thin band of tissue near the superior medial edge of the vocal fold. The cord-like appearance of the ligament gave rise to the traditional term "vocal cord". The ligament connects the arytenoid cartilage (lower broad dark region) to the anterior portion of the thyroid cartilage (upper dark region). The slightly thickened endpoints are known as the anterior and posterior macula flava. In the medial-lateral direction, the vocal ligament comprises the intermediate and deep layer of the lamina propria.

The physiological functions of the vocal ligament are not fully understood. One function is to limit mechanical strain (elongation), a general function of most ligaments in the body. A second function may be to produce a firm closure of the glottis by forming a straight edge along the membranous (vibrating) portion of the vocal fold. A strong ligament that can be tensed with exercise is likely to help straighten the edge of the folds. Vocal fold bowing, for example, is a pathological condition often associated with advanced age, but it can also occur in young adults who press their arytenoid cartilages together excessively in speech. Atrophy of the thyroarytenoid muscle, which lies lateral to the ligament, causes the middle of the membranous vocal fold to be retracted from the midline of the glottis. The result is a weak voice because airflow cannot be suddenly shut off for efficient acoustic excitation of the vocal tract. For self-sustained vocal fold vibration, the superficial layer must be very pliable and deformable for mucosal surface-wave motion. The role of the ligament is then to stabilize the vertical motion when large pressures are applied to vocal fold surfaces. The most important known function of the ligament, however, is to widen the fundamental frequency range. The stiffer the ligament, the greater the likelihood that several octaves of fo range can be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years or older
* no current voice disorder
* no history of performance or professional vocal training

Exclusion Criteria:

* history of head/neck cancer, laryngeal surgery, current voice disorder requiring medical management
* cognitive limitations that would prevent them from successfully and safely participating in the study.
* history of gastrointestinal disease or surgery w
* no known neurological or structural abnormalities of vocal folds
* previous laryngeal surgeries;
* allergies to local anesthetics (used to suppress a sensitive gag reflex during laryngeal endoscopic examination);
* cardiac abnormalities;
* recent history of smoking (must be completely smoke-free for six months prior to study commencement because of the effect of smoking on the voice and laryngopharyngeal reflux severity).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Voice Range Profile (VRP) | pre-intervention (initial evaluation)
  a thorough voice range profile will be created by testing the participants lowest (minimum) and highest (maximum) achievable pitches across a spectrum of vocal intensities (soft, medium and loud).
Voice Range Profile (VRP) | 8 weeks post intervention
  a thorough voice range profile will be created by testing the participants lowest (minimum) and highest (maximum) achievable pitches across a spectrum of vocal intensities (soft, medium and loud).
Voice Range Profile (VRP) | 3 months following intervention
  a thorough voice range profile will be created by testing the participants lowest (minimum) and highest (maximum) achievable pitches across a spectrum of vocal intensities (soft, medium and loud).

SECONDARY OUTCOMES:
Electroglottography (EGG) | pre-intervention
  Electroglottograph, or EGG, is a device used for the noninvasive measurement of the degree of contact between the vibrating vocal folds during voice production. Electrodes are applied on the surface of the neck so that the EGG records variations in the transverse electrical impedance of the larynx can be measured.
Electroglottography (EGG) | 8 weeks post intervention
  Electroglottograph, or EGG, is a device used for the noninvasive measurement of the degree of contact between the vibrating vocal folds during voice production. Electrodes are applied on the surface of the neck so that the EGG records variations in the transverse electrical impedance of the larynx can be measured.
Electroglottography (EGG) | 3 months following treatment.
  Electroglottograph, or EGG, is a device used for the noninvasive measurement of the degree of contact between the vibrating vocal folds during voice production. Electrodes are applied on the surface of the neck so that the EGG records variations in the transverse electrical impedance of the larynx can be measured.
Acoustic measurement | pre-intervention
  An audio recording of each participant will be obtained. The participant will sustain the "ah" and "ee" vowel three times for the maximum amount of time they are able. They will then read the CAPE-V (Zraick et al., 2011), rainbow passage (Fairbanks, 1960), and describe the cookie theft picture (Borod et al., Boston Diagnostic Aphasia Examination 1980). The samples will then be analyzed using Phonanium, an automated acoustic analysis software. Acoustics will include fundamental frequency, fundamental frequency standard deviation, relative sound pressure level (SPL), SPL standard deviation, cepstral peak prominence smooth (CPPS), harmonic to noise ratio, and noise to harmonic ratio, acoustic voice quality index (AVQI), and spectral slope.
Acoustic measurement | 8 weeks post intervention
  An audio recording of each participant will be obtained. The participant will sustain the "ah" and "ee" vowel three times for the maximum amount of time they are able. They will then read the CAPE-V (Zraick et al., 2011), rainbow passage (Fairbanks, 1960), and describe the cookie theft picture (Borod et al., Boston Diagnostic Aphasia Examination 1980). The samples will then be analyzed using Phonanium, an automated acoustic analysis software. Acoustics will include fundamental frequency, fundamental frequency standard deviation, relative sound pressure level (SPL), SPL standard deviation, cepstral peak prominence smooth (CPPS), harmonic to noise ratio, and noise to harmonic ratio, acoustic voice quality index (AVQI), and spectral slope.
Acoustic measurement | 3 months following treatment.
  An audio recording of each participant will be obtained. The participant will sustain the "ah" and "ee" vowel three times for the maximum amount of time they are able. They will then read the CAPE-V (Zraick et al., 2011), rainbow passage (Fairbanks, 1960), and describe the cookie theft picture (Borod et al., Boston Diagnostic Aphasia Examination 1980). The samples will then be analyzed using Phonanium, an automated acoustic analysis software. Acoustics will include fundamental frequency, fundamental frequency standard deviation, relative sound pressure level (SPL), SPL standard deviation, cepstral peak prominence smooth (CPPS), harmonic to noise ratio, and noise to harmonic ratio, acoustic voice quality index (AVQI), and spectral slope.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Maxfield, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No